CLINICAL TRIAL: NCT03342339
Title: Influence of Emotions on Decision-making in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1708168; 2017-A02690-53 (Other: ANSM)
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: influence of emotions; positif emotional induction; decision making; Iowa Gambling Task
MeSH Terms: conditions — Parkinson Disease | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with Parkinson's disease (Other): 1. cognitive examination : mini mental test of Parkinson, Hospital Anxiety and Depression Scale, 5 words by Dubois, fast test frontal assessment, Trail Making Test
  2. viewing of video : scale of differential emotions and Positive and Negative Affect Scale
  3. Test of Iowa Gambling Task
  Interventions: Other: cognitive examination; Other: viewing of video; Other: Iowa Gambling Task
- witnesses (Other): 1. cognitive examination : mini mental test of Parkinson, Hospital Anxiety and Depression Scale, 5 words by Dubois, fast test frontal assessment, Trail Making Test
  2. viewing of video : scale of differential emotions and Positive and Negative Affect Scale
  3. Test of Iowa Gambling Task
  Interventions: Other: cognitive examination; Other: viewing of video; Other: Iowa Gambling Task

INTERVENTIONS:
Other: cognitive examination — mini mental test of Parkinson, Hospital Anxiety and Depression Scale, 5 words by Dubois, fast test frontal assessment, Trail Making Test
Other: viewing of video — viewing during 5 minutes scale of differential emotions and Positive and Negative Affect Scale
Other: Iowa Gambling Task — Test of Iowa Gambling Task

SUMMARY:
Parkinson's disease mainly affects the dopaminergic neurons of the Substancia nigra, which project on the striatum. Neuronal death within this structure leads to a decrease in dopamine levels. Dopamine is a neurotransmitter essential to the proper functioning of the basal ganglia highly involved in the control of voluntary and involuntary movements.

It also leads to cognitive and behavioral changes. Among these changes, the investigators will mainly remember the idea of the emergence of difficulties to make the right decisions, for example at the financial, medical .... This disruption would be the result of executive dysfunction. By definition, executive functions allow us to evaluate, plan and organize our actions to achieve a goal.

DETAILED DESCRIPTION:
Some research shows that positive emotional states are associated with greater self-confidence, greater optimism, and better regulation of our decision-making. The goal is to test whether positive emotional induction could improve decision-making in Parkinson's disease.

Listening to music would decrease anxiety levels and increase self-esteem levels. Who says Parkinson says dopamine deficiency and so the investigators can think that the investigators can help patients by inducing a positive emotion through musical stimulation.

All participants will be subject to emotional induction. They will be divided into two different conditions: either they will be induced in a positive state, or they will be maintained in a neutral state. For this, video clips (positive or neutral) containing music will be presented. Immediately after the presentation of the video, participants will have to perform the Iowa Gambling Task test. This is a sequential task to evaluate decision-making capabilities.

ELIGIBILITY:
Inclusion Criteria for patients :

* Diagnosis of the disease carried out by a hospital doctor
* Stable treatment for two months minimum.
* Mini-Mental Parkinson > 26
* Under dopaminergic treatment

Exclusion Criteria for patients :

* other neurological or psychiatric antecedents
* anxio-depressive symptomatology
* delusional or psychotic state

Inclusion Criteria for witnesses :

* matched in age and sex
* Vision and hearing normal or successfully corrected
* Understand the French language
* general level in the test standard

Exclusion Criteria for witnesses :

* neurological or psychiatric diseases
* anxio-depressive symptomatology

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
net score of Iowa Gambling Task Test | day 1
  calculated by adding the number of cards taken in the right pile and subtracting it from the number of cards chosen in the wrong pile

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Grenoble Alpes, Grenoble
  - CHU de Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No